CLINICAL TRIAL: NCT06103474
Title: Clinical Reporting to Alleviate the Nocebo Effect (CRANE)
Brief Title: Clinical Reporting to Alleviate the Nocebo Effect
Acronym: CRANE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: American Roentgen Ray Society (Other)
Responsible Party: Principal Investigator, Steven A Rothenberg, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 300010891; 000538053 (Other Grant/Funding Number: American Roentgen Ray Society)
Record Dates: First submitted 2023-10-18; First posted 2023-10-26 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Nocebo Effect

STUDY DESIGN:
Intervention Model Description: Survey, cross-sectional study of sixty (n=60) participants undergoing MRI for lower back pain will be randomized to receive an anatomic report (standard of care) versus a Clinical Report (CR). Ordering physicians receiving the Clinical Reports will be instructed to avoid terms that may result in cyberchondria or fear (e.g. disc bulge or nerve impingement) when discussing MRI results.
Who Masked: Investigator
Masking Description: Interpreting radiologists will be blinded to survey data. The PI will be blinded to the intervention type during the review.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Standard of Care Report (Active Comparator): The subject will receive standard of care imaging report.
  Interventions: Diagnostic Test: Lumbar Magnetic Resonance Imaging (MRI)
- Clinical Report (Active Comparator): The subject will receive a technical report that avoids language that may cause catastrophizing or evoke the nocebo effect.
  Interventions: Diagnostic Test: Lumbar Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Diagnostic Test: Lumbar Magnetic Resonance Imaging (MRI) — Lumbar Magnetic Resonance Imaging (MRI)

SUMMARY:
Terminology in radiology reports may cause patients harm by anchoring to or justifying a particular diagnosis. This phenomenon is known as the nocebo effect. MRI may cause patients to pursue more invasive procedures with little added benefit. This study aims to reproduce a study to determine the impact of clinical reporting on patient care and outcomes for those suffering from lower back pain.

ELIGIBILITY:
Inclusion Criteria:

* History of lower back pain undergoing MRI
* Greater than 18 years of age
* Able to understand and willing to comply with all study procedures and is available for the duration of the study

Exclusion Criteria:

* A potential subject who meets any of the following criteria will be excluded from participation in the study:

  * Acute lower back pain secondary to trauma within 1 months
  * Severe cord compression on MRI
  * Cord signal abnormality on MRI
  * Metastatic cancer
  * Spinal epidural abscess
  * Vertebral osteomyelitis
  * Judgement of the ordering physician (e.g. focal neurologic deficit)
  * Anything that, in the opinion of the investigator or team, would place the subject at increased risk or preclude the subject's full compliance with or completion of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2024-01-14 (Actual); Primary Completion 2025-11-11 (Actual); Study Completion 2025-11-11 (Actual)

PRIMARY OUTCOMES:
Improvement of the visual analog scale (VAS) pain score in Clinical Report Cohort. | 6 weeks post intervention
Improvement of the visual analog scale (VAS) pain score in Clinical Report Cohort. | within 7 days post intervention

SECONDARY OUTCOMES:
Improvement in pain interference measured via brief pain inventory | 6 weeks post intervention

CONTACTS AND LOCATIONS:
Locations (1):
- UAB, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No